CLINICAL TRIAL: NCT06893367
Title: Reliability of Sensor-Derived Measurements of the SENSorized Fugl-Meyer (FMA) in Subjects with Stroke Outcomes
Acronym: FMA-SENS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: University of Florence (Other); University of Bucharest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FMA-SENS
Record Dates: First submitted 2025-03-06; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Sensorimotor Impairment Affecting the Upper Limb; 18 Years and Over
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stroke group (Experimental): each participant will perform the FMA with IMU
  Interventions: Device: IMU and RealSense Cameras

INTERVENTIONS:
Device: IMU and RealSense Cameras — Each participant will perform the FMA-sens, with their most affected hand, followed by the FMA-sens with the less affected hand.

SUMMARY:
This study will be conducted at a single research center, the main objective of the study will be to evaluate the efficacy, safety, and accuracy of a medical device that has not yet been commercialized; therefore, it is still under development or testing and is not yet available for private use and is not for profit (nonprofit).

Fifty participants will be recruited from subjects afferent to the outpatient and inpatient neuro-motor rehabilitation clinics of IRCCS Fondazione Don Carlo Gnocchi in Florence, Italy, and afferent to the outpatient and inpatient rehabilitation clinics of Elias University Emergency Hospital in Bucharest, Romania.

In detail, it is deemed necessary to collect clinical and instrumental data. The study will be conducted by an interdisciplinary team composed of healthcare professionals and engineers afferent to the Department of Industrial Engineering.

Should you decide to participate in the study, a visit to verify the inclusion and exclusion criteria will be primarily conducted. Once the admission criteria have been verified, participants will undergo a series of assessments.

The first, involves the administration of some specific sections of the Fugl-Meyer scale (FMA), focusing on the upper extremities. Specifically, the following will be examined: section A for general upper limb function, section B assessing wrist mobility, and finally section D for limb coordination and speed.

During this phase, both upper limbs will be assessed, in addition, the first examiner will carefully place sensors on the participants and assign scores to the tests performed, according to the criteria established by the FMA scale.

Next, a second assessment (T1) will be conducted, in which a second examiner will be responsible for placing the sensors and recording data only on the most affected side.

At a third time, called "T2" and again with at least 15 minutes interval from T1, the first examiner will repeat the same assessments performed in "T1." While performing these assessments, a RealSense camera will be used.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older;
* stroke outcomes with the presence of sensorimotor impairment in the upper limb;
* willingness to participate in the project, with informed consent signed by the person himself or, when necessary, by the support administrator/legal guardian.

Exclusion Criteria:

* Severe concomitant pathologies that modify the subject's motor framework;
* severe visual and/or hearing impairments that cannot be corrected;
* severe neuropsychological impairments (aphasia, apraxia, other cognitive deficits ) such as to prevent cooperation in administering the scale;
* presence of signs of clinical instability, defined by a score greater than zero on the SIC scale (Clinical Instability Scale).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Participants assessed by IMU | baseline
  The Fugl-Meyer Assessment (FMA) is obtained with IMU and RealSense cameras.
  Below are the individual items of the FMA that will be acquired via the experimental kit:
  * A II. Voluntary movement in synergy: flexor synergy/extensor synergy
  * A III. Voluntary movement with mixed synergies: hand to lumbar spine/shoulder flexion 0- 90/pronation-supination
  * A IV. Voluntary movement with reduced or absent synergy: shoulder abduction 0-90/shoulder flexion 90-180/pronation-supination
  * B I. Wrist: stability at 15° dorsiflexion with elbow 90°
  * B II. Wrist: repeated dorsiflexion with elbow 90°
  * B III. Wrist: Stability at 15° dorsiflexion with elbow at 0°
  * B IV. Wrist: repeated dorsiflexion with elbow at 0°
  * D. Coordination/Speed: tremor
  * D. Coordination/Speed: dysmetria
  * D. Coordination/Speed: time
Participants assessed by IMU | at least 15 min from baseline
  The Fugl-Meyer Assessment (FMA) is obtained with IMU and RealSense cameras.
  Below are the individual items of the FMA that will be acquired via the experimental kit:
  * A II. Voluntary movement in synergy: flexor synergy/extensor synergy
  * A III. Voluntary movement with mixed synergies: hand to lumbar spine/shoulder flexion 0- 90/pronation-supination
  * A IV. Voluntary movement with reduced or absent synergy: shoulder abduction 0-90/shoulder flexion 90-180/pronation-supination
  * B I. Wrist: stability at 15° dorsiflexion with elbow 90°
  * B II. Wrist: repeated dorsiflexion with elbow 90°
  * B III. Wrist: Stability at 15° dorsiflexion with elbow at 0°
  * B IV. Wrist: repeated dorsiflexion with elbow at 0°
  * D. Coordination/Speed: tremor
  * D. Coordination/Speed: dysmetria
  * D. Coordination/Speed: time
Participants assessed by IMU | at least 30 min from baseline
  The Fugl-Meyer Assessment (FMA) is obtained with IMU and RealSense cameras.
  Below are the individual items of the FMA that will be acquired via the experimental kit:
  * A II. Voluntary movement in synergy: flexor synergy/extensor synergy
  * A III. Voluntary movement with mixed synergies: hand to lumbar spine/shoulder flexion 0- 90/pronation-supination
  * A IV. Voluntary movement with reduced or absent synergy: shoulder abduction 0-90/shoulder flexion 90-180/pronation-supination
  * B I. Wrist: stability at 15° dorsiflexion with elbow 90°
  * B II. Wrist: repeated dorsiflexion with elbow 90°
  * B III. Wrist: Stability at 15° dorsiflexion with elbow at 0°
  * B IV. Wrist: repeated dorsiflexion with elbow at 0°
  * D. Coordination/Speed: tremor
  * D. Coordination/Speed: dysmetria
  * D. Coordination/Speed: time

SECONDARY OUTCOMES:
Total FMA score | baseline
  Sensorimotor recovery assessment after stroke, total score from 0 to 64, subscore upper limb 36, lower limb 28. Higher scores represent better outcomes.
MODIFIED BARTHEL INDEX (mBI) | baseline
  The Modified Barthel Index (MBI) is a tool used to assess a person's level of independence in performing activities of daily living, particularly in geriatrics and rehabilitation settings. It consists of 10 activities, such as eating, dressing, using the bathroom, moving around, and personal hygiene, each assigned a specific score. A higher score indicates greater independence, while a lower score reflects a higher level of dependence on assistance. The modified version of the Barthel Index is adapted from the original and is commonly used to track progress during rehabilitation or for patients with disabilities.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Firenze, Florence, Italy